CLINICAL TRIAL: NCT04628182
Title: The China Laparoscopic Right Hemicolectomy SNAPSHOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Other Study IDs: BFH SNAPSHOT
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Right Hemicolectomy; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to explore the current practice of right hemicolectomy for colon cancer located in the ascending colon and hepatic flexure in selected Chinese high quality and high volume centres. This study will identify a potential area to improve the level of standard care and serve as a reference cohort to which planned standardization and addition of innovative aspects can be compared to

ELIGIBILITY:
Inclusion Criteria:

* Segmental right sided hemicolectomy (including extended)
* Cancer stage 1-3 (CT-staged)
* No prior abdominal surgery

Exclusion Criteria:

* Stage cT4b, perforated disease
* Acute obstruction
* Emergency surgery
* Right hemicolectomy or ileocaecal resection as part of a large procedure such as subtotal colectomy or panproctocolectomy
* Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with non-metastasized right sided colon cancer without ingrowth into other organs suitable for elective radical resection of the ascending colon.
Sampling Method: Non-Probability Sample
Enrollment: 1579 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
post-operative anastomotic leakages | 1 month
  Number of post-operative anastomotic leakages within 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China